CLINICAL TRIAL: NCT00230594
Title: Desmopressin Response in the Young: A Double-blind, Randomised, Placebo-controlled, Dose-titration Study With Three Different Doses (120 Mcg, 240 Mcg and 360 Mcg) of Desmopressin Administered as a New Melt Tablet in Children and Adolescents With Primary Nocturnal Enuresis (PNE).
Brief Title: Desmopressin Response in the Young
Acronym: DRY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FE992026, CLN 10.3.26
Record Dates: First submitted 2005-09-28; First posted 2005-10-03 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Primary Nocturnal Enuresis
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): desmopressin
  Interventions: Drug: desmopressin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desmopressin — desmopressin 120 mcg melt tablet; 120 mcg, 240 mcg or 360 mcg administered once daily before bedtime
  Other Names: DDAVP
  Arms: 1
Drug: placebo — placebo melt tablet; 1 to 3 placebo melt tablets administered once daily before bedtime
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether desmopressin administered as a melt tablet is effective in reducing the number of wet nights in children and adolescents who suffer from bedwetting.

DETAILED DESCRIPTION:
Primary nocturnal enuresis (PNE), or bedwetting, is a common childhood urological disease. Factors contributing to nocturnal enuresis include nocturnal polyuria due to, at least in part, a relative deficiency of antidiuretic hormone arginine vasopressin (AVP) which has been supported by the finding that some enuretic children lack a nocturnal increase in endogenous AVP secretion. Desmopressin, a synthetic, structural analogue of AVP, selective for V2-receptors and with a longer half life than the natural hormone, has been found to be especially beneficial in PNE subjects with nocturnal polyuria and normal functional bladder capacity.

A melt tablet formulation offers benefits compared to regular tablets and nasal spray. Regular tablets are more difficult to swallow for some patients and require fluid intake for swallowing. Nasal spray absorption may be altered by seasonal allergies, upper respiratory infections or improper administration.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (age 5-16 years) with diagnosed primary monosymptomatic nocturnal enuresis.
* A minimum of 3 wet nights per week in the 2-week screening period without treatment.

Exclusion Criteria:

* Presence or a history of organic urological disease, diurnal urinary incontinence, polydipsia, diabetes insipidus, ongoing urinary tract infection, clinically significant renal, hepatic, gastrointestinal, pulmonary, cardiovascular, endocrinological or neurological disease that would interfere with evaluation.
* Ongoing systemic antibiotic use, use of diuretics or any drugs affecting urinary concentration, or medical treatment for hyperactivity.
* Usage of any experimental drug or device during 30 days before study entry.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2004-07; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of desmopressin administered as a melt tablet compared to placebo in terms of reducing the number of wet nights in children and adolescents with primary nocturnal enuresis. | 14 days of screening plus 54 days of treatment

SECONDARY OUTCOMES:
To evaluate the efficacy of desmopressin administered as a melt tablet compared to placebo in terms of percentage baseline reduction in the number of wet nights. | 14 days of screening plus 54 days of treatment
To evaluate the efficacy of desmopressin administered as a melt tablet compared to placebo in terms of the proportion of full, partial and non-responders. | 14 days of screening plus 54 days of treatment
To investigate the safety and tolerability of desmopressin, administered as a melt tablet compared to placebo, for all doses tested. | 14 days of screening plus 54 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (9):
- Canada (9):
  - IWK Health Centre, Halifax, Nova Scotia
  - The Male Health Centres, Barrie, Ontario
  - Cambridge Family Medical Centre, Cambridge, Ontario
  - Private Clinic, London, Ontario
  - Quest Clinical Trials Inc., Markham, Ontario
  - Private Clinic, North Bay, Ontario
  - The Male Health Centres, Oakville, Ontario
  - Markham Place Med Centre, Thornhill, Ontario
  - The Kids Clinic, Whitby, Ontario

REFERENCES:
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251